CLINICAL TRIAL: NCT06006624
Title: Single-Shot Liposomal Bupivacaine vs. Liposomal Bupivacaine Combined With Dexamethasone Following Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Controlled Trial
Brief Title: Exparel vs Block for ACL Reconstruction
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHAM2023-2163
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: ACL; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: ACL repair + Exparel + nerve block (Active Comparator): 30 mL Liposomal bupivacaine (Exparel) + 5 cc's of 0.5% bupivacaine evenly distributed and administered in adductor canal and iPACK block (35 mL total)
  Interventions: Drug: Exparel 30 mL; Drug: 0.5% bupivacaine; Drug: iPACK block
- Group 2: ACL repair + Exparel + Dexamethasone + nerve block (Active Comparator): 30 mL Liposomal bupivacaine (Exparel) + 10 mg preservative free Dexamethasone + 5 cc's of 0.5% bupivacaine evenly distributed for both adductor canal and iPACK block (35 mL total)
  Interventions: Drug: Exparel 30 mL; Drug: 0.5% bupivacaine; Drug: Dexamethasone; Drug: iPACK block

INTERVENTIONS:
Drug: Exparel 30 mL — 30 mL Liposomal bupivacaine (Exparel) evenly distributed and administered in adductor canal block
Drug: 0.5% bupivacaine — 5 cc's of 0.5% bupivacaine evenly distributed and administered in adductor canal
Drug: Dexamethasone — 10 mg preservative free Dexamethasone evenly distributed and administered in adductor canal
  Arms: Group 2: ACL repair + Exparel + Dexamethasone + nerve block
Drug: iPACK block — iPACK (Infiltration between the Popliteal artery and Capsule of the Knee) block

SUMMARY:
Liposomal bupivacaine or Exparel (Pacira Biosciences) is a long-lasting nonopioid analgesic that was initially utilized as an infiltrative agent but has more recently become U.S. Food and Drug Administration (FDA) approved for use in interscalene brachial plexus nerve blockade as well as infiltrative blockade. Delivery in this form is reported to provide up to 72 hours of extended-release bupivacaine. Exparel's use as a regional anesthetic has also become increasingly common and has shown promise when utilized in Anterior Cruciate Ligament (ACL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Paticipants with ACL rupture amenable to reconstruction with BTB autograft identified in clinic by one of 4 different surgeons
* Primary ACL Reconstruction with Autograft +/- Partial meniscectomy +/- Lateral extra-articular tenodesis
* Age 18 and older
* English speaking
* Ability to complete surveys by phone or in person
* Ability to provide informed consent

Exclusion Criteria:

* Revision cases
* Multi-ligamentous knee injuries
* Cartilage or meniscal procedures that prevent adherence to immediate weight bearing and range of motion rehab protocol
* ACL reconstruction utilizing non-bone-patellar tendon-bone autografts
* Allergies to study medications
* Non-English speakers
* Known alcohol or narcotic abuse history
* Existing contract with a pain specialist due to underlying preoperative pain syndrome
* Preoperative opioid use within the 3 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 14 days
  Daily postoperative VAS (visual analog scale for pain) scale will be collected from participants to assess pain
Postoperative opioid use | 14 days
  assessed using a participant daily diary of how much medication was taken daily for pain
Postoperative Pain #2 | 14 days
  Daily postoperative NRS (numerical rating scale for pain) scale will be collected from participants to assess pain

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Johns WL, Voskeridjian A, Miltenberg B, Muchintala R, Dodson CC, Cohen SB, Salvo J, Sherman M, Ciccotti MG, Hammoud S. Regional Anesthesia Utilizing Liposomal Bupivacaine, With or Without Dexamethasone, Provides Excellent Pain Control and Minimizes Opioid Consumption Following Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2026 Jan 8;14(1):23259671251401596. doi: 10.1177/23259671251401596. eCollection 2026 Jan. PMID 41522461